CLINICAL TRIAL: NCT04537793
Title: A Phase 3 Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Elexacaftor/Tezacaftor/Ivacaftor Triple Combination Therapy in Cystic Fibrosis Subjects 2 Through 5 Years of Age
Brief Title: Evaluation of ELX/TEZ/IVA in Cystic Fibrosis (CF) Subjects 2 Through 5 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VX20-445-111; 2020-002251-38 (EudraCT Number)
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: ELX/TEZ/IVA (Experimental): Participants weighing greater than or equal to (>=)14 kilograms (kg) at screening received elexacaftor (ELX) 100 milligrams (mg) once daily (qd)/tezacaftor (TEZ) 50 mg qd/ivacaftor (IVA) 75 mg every 12 hours (q12h) in the treatment period for 15 days.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA
- Part B: ELX/TEZ/IVA (Experimental): Participants weighing (>=)14 kg at screening received ELX 100 mg qd/TEZ 50 mg qd/IVA 75 mg q12h. Participants weighing (>=)10 kg to less than (<)14 kg received ELX 80 mg qd/TEZ 40 mg qd/IVA 60 mg once every morning (qAM) and 59.5 mg once every evening (qPM) in the treatment period for 24 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed dose combination granules for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
Drug: IVA — Granules for oral administration.
  Other Names: VX-770; ivacaftor

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy of elexacaftor (ELX)/tezacaftor (TEZ)/ivacaftor (IVA) triple combination therapy in CF subjects 2 through 5 years of age.

ELIGIBILITY:
Key Inclusion Criteria:

* Homozygous for the F508del mutation or heterozygous for F508del and a minimal function (MF) mutation (F/F or F/MF genotypes)

Key Exclusion Criteria:

* Clinically significant cirrhosis with or without portal hypertension
* Lung infection with organisms associated with a more rapid decline in pulmonary status
* Solid organ or hematological transplantation

Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (13):
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Stanford University, Palo Alto, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Respiratory and Critical Care Specialists, P.A., Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine / St. Louis Children's Hospital, St Louis, Missouri
  - NC TraCS Institute - CTRC University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
- Australia (3):
  - Telethon Kids Institute, Nedlands
  - The Royal Children's Hospital, Parkville, VIC
  - Queensland Children's Hospital, South Brisbane
- Canada (2):
  - The Hospital for Sick Children, Toronto
  - British Columbia Children's Hospital, Vancouver
- Germany (2):
  - Charite Paediatric Pulmonology Department, Berlin
  - Universitatsklinikum Essen (AoR), Kinderklinik III, Abt. fur Pneumologie, Essen
- United Kingdom (2):
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Goralski JL, Hoppe JE, Mall MA, McColley SA, McKone E, Ramsey B, Rayment JH, Robinson P, Stehling F, Taylor-Cousar JL, Tullis E, Ahluwalia N, Chin A, Chu C, Lu M, Niu T, Weinstock T, Ratjen F, Rosenfeld M. Phase 3 Open-Label Clinical Trial of Elexacaftor/Tezacaftor/Ivacaftor in Children Aged 2-5 Years with Cystic Fibrosis and at Least One F508del Allele. Am J Respir Crit Care Med. 2023 Jul 1;208(1):59-67. doi: 10.1164/rccm.202301-0084OC. PMID 36921081
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 parts, Part A and Part B. The Participant flow was planned to be presented for the overall treatment arms (i.e. Part A and Part B), irrespective of weight-based dose regimen.
Pre-assignment Details: This study was conducted in participants with cystic fibrosis (CF) aged 2 through 5 years of age (inclusive).
Groups:
- Part A: ELX/TEZ/IVA: Participants weighing greater than or equals to (>=)14 kg at screening received elexacaftor (ELX) 100 milligrams (mg) once daily (qd)/tezacaftor (TEZ) 50 mg qd/ivacaftor (IVA) 75 mg every 12 hours (q12h) in the treatment period for 15 days.
- Part B: ELX/TEZ/IVA: Participants weighing >=14 kg at screening received ELX 100mg qd/TEZ 50mg qd/IVA 75 mg q12h and participants weighing >=10 kg to less than (<)14 kg received ELX 80mg qd/TEZ 40mg qd/IVA 60 mg once every morning (qAM) and IVA 59.5 mg once every evening (qPM) in the treatment period for 24 weeks.
Period: Part A (15 Days)
Arm/Group | Part A: ELX/TEZ/IVA | Part B: ELX/TEZ/IVA
Started | 18 | 0
Completed | 18 | 0
Not Completed | 0 | 0
Period: Part B (24 Weeks)
Arm/Group | Part A: ELX/TEZ/IVA | Part B: ELX/TEZ/IVA
Started | 0 | 75 (Out of the 18 participants from Part A, 10 participants also participated in Part B of the study.)
Completed | 0 | 74
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug during the treatment period were included in the baseline analysis.
Groups:
- ELX/TEZ/IVA: Part A: Participants weighing greater than or equal to (>=)14 kilograms (kg) at screening received ELX 100 milligrams (mg) once daily (qd)/TEZ 50 mg qd/IVA 75 mg every 12 hours (q12h) in the treatment period for 15 days.
  Part B: Participants weighing >=14 kg at screening received ELX 100mg qd/TEZ 50mg qd/IVA 75 mg q12h and participants weighing >=10 kg to less than (<)14 kg received ELX 80mg qd/TEZ 40mg qd/IVA 60 mg once every morning (qAM) and IVA 59.5 mg once every evening (qPM) in the treatment period for 24 weeks.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 83
Age, Categorical [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented for the overall treatment arms (i.e. Part A and Part B), irrespective of weight-based dose regimen. Here "number analyzed" signifies participants who were evaluable for specified part of the study.
  Participants
    Part A: number analyzed (Participants) | 18
    Part A: <=18 years | 18
    Part A: Between 18 and 65 years | 0
    Part A: >=65 years | 0
    Part B: number analyzed (Participants) | 75
    Part B: <=18 years | 75
    Part B: Between 18 and 65 years | 0
    Part B: >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented for the overall treatment arms (i.e. Part A and Part B), irrespective of weight-based dose regimen. Here "number analyzed" signifies participants who were evaluable for specified part of the study.
  Participants
    Part A: number analyzed (Participants) | 18
    Part A: Female | 11
    Part A: Male | 7
    Part B: number analyzed (Participants) | 75
    Part B: Female | 41
    Part B: Male | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented for the overall treatment arms (i.e. Part A and Part B), irrespective of weight-based dose regimen. Here "number analyzed" signifies participants who were evaluable for specified part of the study.
  Participants
    Part A: number analyzed (Participants) | 18
    Part A: Hispanic or Latino | 0
    Part A: Not Hispanic or Latino | 18
    Part A: Not collected per local regulations | 0
    Part B: number analyzed (Participants) | 75
    Part B: Hispanic or Latino | 6
    Part B: Not Hispanic or Latino | 63
    Part B: Not collected per local regulations | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented for the overall treatment arms (i.e. Part A and Part B), irrespective of weight-based dose regimen. Here "number analyzed" signifies participants who were evaluable for specified part of the study.
  Participants
    Part A: number analyzed (Participants) | 18
    Part A: White | 18
    Part A: Black or African American | 0
    Part A: Not collected per local regulations | 0
    Part B: number analyzed (Participants) | 75
    Part B: White | 68
    Part B: Black or African American | 1
    Part B: Not collected per local regulations | 6

OUTCOME MEASURES:

1. Primary Outcome: Part A: Observed Pre-dose Concentration (Ctrough) of ELX,TEZ,IVA, and Relevant Metabolites
Time Frame: From Day 1 through Day 15
Population: Pharmacokinetic (PK) set included participants who received at least 1 dose of study drug. Here the "Number Analyzed" signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/ml)
Groups:
- Part A: ELX/TEZ/IVA: Participants weighing >=14 kg at screening received ELX 100 mg qd/TEZ 50 mg qd/IVA 75 mg q12h in the treatment period for 15 days.
Arm/Group | Part A: ELX/TEZ/IVA
Number analyzed (Participants) | 18
micrograms per milliliter (mcg/ml)
  Day 1: ELX | 0.00 (0.00)
  Day 8: ELX | 3.44 (2.09)
  Day 15: ELX: number analyzed (Participants) | 17
  Day 15: ELX | 3.69 (2.11)
  Day 1: ELX-M23 | 0.00 (0.00)
  Day 8: ELX-M23 | 2.39 (1.65)
  Day 15: ELX-M23: number analyzed (Participants) | 17
  Day 15: ELX-M23 | 2.47 (1.65)
  Day 1: TEZ | 0.00 (0.00)
  Day 8: TEZ | 1.86 (1.07)
  Day 15: TEZ: number analyzed (Participants) | 17
  Day 15: TEZ | 1.85 (1.10)
  Day 1: TEZ-M1 | 0.00 (0.00)
  Day 8: TEZ-M1 | 6.42 (1.42)
  Day 15: TEZ-M1: number analyzed (Participants) | 17
  Day 15: TEZ-M1 | 7.68 (1.52)
  Day 1: IVA | 0.00 (0.00)
  Day 8: IVA | 0.702 (0.503)
  Day 15: IVA: number analyzed (Participants) | 17
  Day 15: IVA | 0.746 (0.526)
  Day 1: IVA-M1 | 0.00 (0.00)
  Day 8: IVA-M1 | 1.78 (0.990)
  Day 15: IVA-M1: number analyzed (Participants) | 17
  Day 15: IVA-M1 | 1.91 (0.990)

2. Primary Outcome: Part A: Safety and Tolerability as Assessed by Number of Participants With Treatment- Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From Day 1 up to Day 43
Population: Safety set for Part A included all participants who received at least 1 dose of study drug in Part A. This outcome measure was planned only for Part A arm.
Measure: Number; unit: participants
Arm/Group | Part A: ELX/TEZ/IVA
Number analyzed (Participants) | 18
participants
  Participants with TEAEs | 15
  Participants with SAEs | 0

3. Primary Outcome: Part B: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From Day 1 up to Week 28
Population: Safety set for Part B included all participants who received at least 1 dose of study drug in Part B. The safety and tolerability analysis for Part B was assessed for the overall treatment arm, irrespective of weight-based dose regimen. Therefore, the analysis is reported for the single triple combination (Part B: ELX/TEZ/IVA) arm.
Measure: Number; unit: participants
Groups:
- Part B: ELX/TEZ/IVA: Participants weighing >=14 kg at screening received ELX 100mg qd/TEZ 50mg qd/IVA 75 mg q12h and participants weighing >=10 kg to <14 kg received ELX 80mg qd/TEZ 40mg qd/IVA 60 mg qAM and IVA 59.5 mg qPM in the treatment period for 24 weeks.
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 75
participants
  Participants with TEAEs | 74
  Participants with SAEs | 2

4. Secondary Outcome: Part B: Observed Pre-dose Plasma Concentration (Ctrough) of ELX,TEZ,IVA and Relevant Metabolites
Time Frame: From Day 1 through Week 16
Population: PK set included participants who received at least 1 dose of study drug. Here the "Number Analyzed" signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/ml)
Groups:
- Part B: ELX/TEZ/IVA (≥10 kg to <14 kg): Participants weighing >=10 kg to l <14 kg received ELX80mg qd/TEZ 40mg qd/IVA 60 mg qAM and IVA 59.5 qPM in the treatment period for 24 weeks.
- Part B: ELX/TEZ/IVA (≥14 kg): Participants weighing >=14 kg at screening received ELX100 mg qd/TEZ 50 mg qd/IVA 75 mg q12h in the treatment period for 24 weeks.
Arm/Group | Part B: ELX/TEZ/IVA (≥10 kg to <14 kg) | Part B: ELX/TEZ/IVA (≥14 kg)
Number analyzed (Participants) | 16 | 59
micrograms per milliliter (mcg/ml)
  Day 15: ELX: number analyzed (Participants) | 14 | 54
  Day 15: ELX | 2.91 (1.38) | 3.87 (2.75)
  Week 4: ELX | 3.13 (1.90) | 3.56 (2.19)
  Week 12: ELX: number analyzed (Participants) | 16 | 56
  Week 12: ELX | 2.48 (1.65) | 3.49 (2.22)
  Week 16: ELX: number analyzed (Participants) | 15 | 58
  Week 16: ELX | 3.01 (1.11) | 3.18 (2.19)
  Day 15: ELX-M23: number analyzed (Participants) | 14 | 54
  Day 15: ELX-M23 | 1.85 (1.12) | 2.33 (1.87)
  Week 4: ELX-M23 | 2.32 (2.01) | 2.22 (1.66)
  Week 12: ELX-M23: number analyzed (Participants) | 16 | 56
  Week 12: ELX-M23 | 1.48 (1.27) | 2.17 (1.69)
  Week 16: ELX-M23: number analyzed (Participants) | 15 | 58
  Week 16: ELX-M23 | 1.73 (0.828) | 1.94 (1.58)
  Day 15: TEZ: number analyzed (Participants) | 14 | 52
  Day 15: TEZ | 1.73 (0.666) | 2.14 (1.72)
  Week 4: TEZ | 1.62 (0.716) | 1.79 (0.947)
  Week 12: TEZ: number analyzed (Participants) | 16 | 56
  Week 12: TEZ | 1.60 (0.951) | 1.76 (1.10)
  Week 16: TEZ: number analyzed (Participants) | 15 | 58
  Week 16: TEZ | 1.52 (0.701) | 1.80 (1.42)
  Day 15: TEZ-M1: number analyzed (Participants) | 14 | 52
  Day 15: TEZ-M1 | 7.07 (1.08) | 7.07 (2.11)
  Week 4: TEZ-M1 | 6.80 (1.64) | 7.09 (2.18)
  Week 12: TEZ-M1: number analyzed (Participants) | 16 | 56
  Week 12: TEZ-M1 | 7.06 (2.37) | 7.18 (2.38)
  Week 16: TEZ-M1: number analyzed (Participants) | 15 | 58
  Week 16: TEZ-M1 | 6.88 (1.94) | 6.95 (2.77)
  Day 15: IVA: number analyzed (Participants) | 14 | 52
  Day 15: IVA | 0.549 (0.373) | 0.661 (0.552)
  Week 4: IVA | 0.535 (0.402) | 0.594 (0.405)
  Week 12: IVA: number analyzed (Participants) | 16 | 56
  Week 12: IVA | 0.383 (0.203) | 0.530 (0.474)
  Week 16: IVA: number analyzed (Participants) | 15 | 58
  Week 16: IVA | 0.483 (0.347) | 0.580 (0.511)
  Day 15: IVA-M1: number analyzed (Participants) | 14 | 52
  Day 15: IVA-M1 | 1.47 (0.969) | 1.67 (0.961)
  Week 4: IVA-M1 | 1.64 (1.29) | 1.52 (0.737)
  Week 12: IVA-M1: number analyzed (Participants) | 16 | 56
  Week 12: IVA-M1 | 1.19 (0.602) | 1.45 (0.907)
  Week 16: IVA-M1: number analyzed (Participants) | 15 | 58
  Week 16: IVA-M1 | 1.24 (0.673) | 1.51 (0.911)

5. Secondary Outcome: Part B: Absolute Change in Sweat Chloride (SwCl)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline through Week 24
Population: FAS (Part B). The efficacy analysis for Part B was assessed for the overall treatment arm, irrespective of weight-based dose regimen. Therefore, the analysis is reported for the single triple combination (Part B: ELX/TEZ/IVA) arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Groups:
- Part B: ELX/TEZ/IVA: Participants weighing >=14 kg received ELX 100mg qd/TEZ 50mg qd/IVA 75 mg q12h and participants weighing >=10 kg to <14 kg received ELX 80mg qd/TEZ 40mg qd/IVA 60 mg qAM and IVA 59.5mg qPM in the treatment period for 24 weeks.
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 75
millimole per liter (mmol/L) | -57.9 [-61.3 to -54.6]

6. Secondary Outcome: Part B: Absolute Change in Lung Clearance Index 2.5 (LCI 2.5)
Description: The LCI2.5 index is the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting values and is calculated by dividing the sum of exhaled tidal breaths (cumulative exhaled volume (CEV)) by simultaneously measured functional residual capacity (FRC). An LCI of 7.5 and below is normal; values greater than 7.5 are abnormal. LCI is able to detect abnormalities in lung function earlier than more traditional modalities such as spirometry.
Time Frame: From Baseline through Week 24
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: index
Groups:
- Part B: ELX/TEZ/IVA: Participants weighing >=14 kg received ELX 100 mg qd/TEZ 50mg qd/IVA 75 mg q12h and participants weighing >=10 kg to less than <14 kg received ELX 80 mg qd/TEZ 40mg qd/IVA 60 mg qAM and IVA 59.5 mg qPM in the treatment period for 24 weeks.
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 63
index | -0.83 [-1.01 to -0.66]

ADVERSE EVENTS:
Time Frame: Day 1 Through Safety Follow-up Visit (up to Day 43 for Part A, up to Week 28 for Part B)
Description: The safety analysis for Part B was assessed for the overall treatment arm, irrespective of weight-based dose regimen.Therefore, the analysis is reported for the single triple combination (Part B: ELX/TEZ/IVA) arm.
  MedDRA version 23.1 applied for Part A, MedDRA version 25.0 applied for Part B.
Groups:
- Part B: ELX/TEZ/IVA: Participants weighing >=14 kg at screening received ELX 100 mg qd/TEZ 50 mg qd/IVA 75 mg q12h and participants weighing >=10 kg to <14 kg received ELX 80 mg qd/TEZ 40 mg qd/IVA 60 mg qAM and IVA 59.5 mg qPM in the treatment period for 24 weeks.
Arm/Group | Part A: ELX/TEZ/IVA | Part B: ELX/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/18 | 2/75
Other Adverse Events (participants affected / at risk) | 15/18 | 71/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: ELX/TEZ/IVA (N=18) | Part B: ELX/TEZ/IVA (N=75)
Anal incontinence (Gastrointestinal disorders) | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: ELX/TEZ/IVA (N=18) | Part B: ELX/TEZ/IVA (N=75)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 5
Abdominal pain (Gastrointestinal disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 0 | 5
Vomiting (Gastrointestinal disorders) | 0 | 21
Pyrexia (General disorders) | 1 | 26
COVID-19 (Infections and infestations) | 0 | 14
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 8
Nasopharyngitis (Infections and infestations) | 0 | 6
Upper respiratory tract infection (Infections and infestations) | 1 | 11
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 8
Aspartate aminotransferase increased (Investigations) | 2 | 4
Gamma-glutamyltransferase increased (Investigations) | 1 | 4
SARS-CoV-2 test positive (Investigations) | 0 | 7
Decreased appetite (Metabolism and nutrition disorders) | 0 | 9
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 7
Product taste abnormal (Product Issues) | 1 | 0
Irritability (Psychiatric disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 46
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 13
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 25
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 12
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT04537793/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT04537793/SAP_001.pdf